CLINICAL TRIAL: NCT06958289
Title: Cryoneurolysis for Spasticity Treatment: Quantifying Long-term Clinical Outcomes and Exploring Mechanisms Within the Central Nervous System
Brief Title: Cryoneurolysis for Spasticity Treatment: Long-term Clinical Outcomes and Mechanisms in the Central Nervous System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sue Peters (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Sue Peters, Assistant Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-126338-105529
Record Dates: First submitted 2025-03-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Spasticity as Sequela of Stroke
Keywords: NIRS; TMS; cryoneurolysis; fNIRS

STUDY DESIGN:
Intervention Model Description: This is a mechanistic study where all participants receive the same intervention and assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Each participant will receive cryoneurolysis which involves the application of extreme cold directly to, or near targeted nerves under ultrasound guidance. This cold causes axonotmesis to occur, thereby completely preventing the treated nerve from propagating any signal. Cryoneurolysis produces an effect called Wallerian degeneration, where the treated nerve's axon is destroyed but the epineurium and perineurium are left intact. Therefore, the axon can regenerate, following the same path as prior to treatment.
  Interventions: Device: Cryoneurolysis

INTERVENTIONS:
Device: Cryoneurolysis — Each participant will receive cryoneurolysis which involves the application of extreme cold directly to, or near targeted nerves under ultrasound guidance. This cold causes axonotmesis to occur, thereby completely preventing the treated nerve from propagating any signal. Cryoneurolysis produces an effect called Wallerian degeneration, where the treated nerve's axon is destroyed but the epineurium and perineurium are left intact. Therefore, the axon can regenerate, following the same path as prior to treatment.

SUMMARY:
Spasticity can make regular daily activities difficult or impossible. Cryoneurolysis is a new technique to treat spasticity that is currently being tested. For this technique, a needle is inserted alongside a nerve implicated in spasticity. The needle then freezes and causes the nerve to break down. The nerve breaking down seems to provide relief for spasticity. The investigators are interested in testing the long-term effects of cryoneurolysis on the function of the brain over six months after treatment. The investigators are testing the brain's function using transcranial magnetic stimulation (TMS) which involves a magnet activating specific parts of the brain that cause muscles to fire; magnetic resonance imaging (MRI) which uses to examine brain structure; functional near-infrared spectroscopy (fNIRS) to examine brain function. The investigators believe that there will be a change in these measures that are related to the long-lasting effects of cryoneurolysis. Cryoneurolysis is not a part of standard care after stroke but is approved in Canada for patients. It has been used extensively in the past for treating pain. TMS is a way of studying how the brain sends signals to muscles to make movement. During these sessions, a researcher will use a magnet to turn on specific neurons in the brain that will cause muscles to contract. The investigators can study the way eyes and muscles respond to better understand how the brain is sending information about moving the body to the muscles. FNIRS is a new way of studying how the brain works. During these sessions, a researcher will fit the participant with a cap that has several lights on it. The light travels through hair, scalp, and skull where it interacts with blood in the brain. By studying the changes in the colour of the blood in the brain, researchers can understand which parts of the brain are active during specific tasks. Magnetic Resonance Imaging (MRI) involves a powerful magnet that takes very detailed pictures of the brain. These images help the investigators to understand how a stroke is related to spasticity. Also, these images are helpful to make the stimulation with TMS more accurate. Study participation will require five visits to the Parkwood Institute Main Building and one visit to St. Joseph's Hospital. The entire study will take place over roughly six months. The investigators are recruiting 25 people with stroke who are eligible for cryoneurolysis to participate in the study.

DETAILED DESCRIPTION:
Spasticity is the result of an overactive stretch reflex after an upper motor neuron injury that results in affected muscles being constantly, involuntarily contracted.1 A failure to treat spasticity can result in contracture - a permanent shortening of the muscle and inert tissues often necessitating surgical intervention.2 There are several treatment options available to those affected by spasticity. Pharmaceutical remedies include diazepam, clonidine, and baclofen, which can be administered orally or intrathecally, and target the GABA-B receptors within the brain and spinal cord to alleviate spasticity.3 Because of the central effects, it is impossible to direct the effects towards specific musculature, making this approach most beneficial for patients with widespread spasticity, especially non-ambulatory patients for whom systemic weakness is less of a concern. For those affected by focal spasticity (spasticity that affects specific regions), there are a number of selective treatments available. By far the most common approach is denervation with botulinum-A neurotoxin. Toxin injections are administered at the neuromuscular junction and act to prevent the release of acetylcholine, thereby reducing the ability of the muscle to fire.4 Botulinum toxin is one of the most potent neurotoxins available but is also one of the most expensive substances on the planet. Since each muscle has many neuromuscular junctions, it is impossible to completely denervate a muscle with this technique. Furthermore, peak effects do not generally endure beyond 90 days and the procedure must be repeated frequently.

Recent developments have led to new treatments for focal spasticity. With ultrasound guidance, clinicians are now able to easily visualize individual nerves, creating a new target for intervention. Chemical neurolysis is a developing technique being performed in a small number of clinics worldwide. The procedure involves the selective injection of a diluted phenol solution into or near motor neurons that innervate muscles implicated in spasticity. Phenol neurolysis has been shown to be effective for relieving spasticity in several locations.5-7 Phenol, however, is not selective to nerves and therefore surrounding tissues and structures are not immune to the injections. Nevertheless, chemical neurolysis has a low incidence of side effects.8,9 Chemical neurolysis is much cheaper than toxin injections, but also must be repeated frequently for long-term spasticity alleviation.10 A second, similar approach is neurolysis by pulsed radiofrequency. While phenol lyses targeted nerves with chemicals, pulsed radiofrequency heats nerves with radio-waves to ablate targeted axons. Radiofrequency ablation has been shown to have a very low incidence of side effects, and reduction in spasticity symptoms has been shown to endure six months.11 Cryoneurolysis, another emerging technique for spasticity management, is more cost effective than other techniques, and the effects outlast the expected effect period.12 Cryoneurolysis involves the application of extreme cold directly to, or near targeted nerves under ultrasound guidance. This cold causes axonotmesis (the breakdown of an axon) to occur, thereby completely preventing the treated nerve from propagating any signal. Taking advantage of the Joule Thomson effect (the cooling of compressed gases with a thin aperture), cryoneurolysis probes are specially designed to quickly create a ball of ice by freezing interstitial fluid. This procedure has been demonstrated to be effective in interventional pain management, by lysing nerves that are involved in the transmission of pain signals.13-18 The investigators have published data showing the effectiveness of cryoneurolysis on spasticity affecting the upper and lower limbs.12,19-21 Cryoneurolysis produces an effect called Wallerian degeneration, where the treated nerve's axon is destroyed but the epineurium and perineurium are left intact.22 Therefore, the axon can regenerate, following the same path as prior to treatment. Preliminary data show that reductions in spasticity from cryoneurolysis endure even after the nerve has regrown, with patients seeing lasting benefits after a full year.12 While the mechanism by which spasticity severity is reduced after cryoneurolysis is a topic of debate in the field, the sustained benefits from the procedure imply central nervous system (CNS) involvement. Our hypothesis is that neuroplastic changes are likely occurring in the CNS that allow for the long-term improvement of spasticity. These changes may be related to changes within the cortex or the output of cortical processing, or some combination of these mechanisms. Thus, the mechanism may involve one or more regions within the cortex and/or changes along the corticospinal tract, the main descending tract that carries movement related information from the CNS to the periphery.

Measuring changes in brain organization and activity have become possible through advances in neuroimaging and stimulation techniques. Transcranial magnetic stimulation (TMS) is a safe, non-invasive method used to stimulate cortical regions to measure levels of cortical excitability, and the output of the processing of information in the cortex through the corticospinal tract. Cortical excitability of the primary motor cortex (M1) is assessed indirectly by measuring electromyographic (EMG) responses (motor evoked potentials; MEPs) of a target motor cortical muscle representation, and brain function is inferred from measurements of peripheral muscle activity. Considerable attention has been paid recently to neuroplastic changes in the brain that occur with interventions. Surface EMG has been used for decades to understand muscle activation patterns. Typically, a pair of electrodes are placed over a muscle group to give an indication of the level of corticospinal excitability that can be telling of the quality and integrity of motor output to the spinal cord.23 This technique provides a look into the output of cortical mechanisms of movement production. The investigators have shown ipsilateral and contralateral changes in cortical excitability of the sensorimotor cortices with TMS in patients with stroke.24 However, after a stroke, if the corticospinal tract has incurred sufficient damage, patients with stroke will not be able to reliably produce an MEP.

While sitting quietly, not completing any active tasks and in the absence of any stimulus, the brain remains active. Resting state functional connectivity (rsFC) is a neuroimaging technique that studies regions of the brain with temporally correlated activation. Longitudinally post stroke, rsFC has been shown to produce similar findings to connectivity analyses in task-based studies;26 however, in contrast to task-based neuroimaging studies, rsFC does not require the participant to be able to move in specific ways and does not have any cognitive demand, thus lowering the burden on participants. Cross-sectional studies of stroke rehabilitation have demonstrated correlations between rsFC and mobility after stroke.27 In spasticity, a 2023 functional magnetic resonance imaging (fMRI) study of spasticity treatment with spinal cord stimulation found that the treatment produced clinical spasticity improvements that correlated with functional connectivity changes.28 The majority of rsFC studies in stroke rehabilitation have been conducted using fMRI. Functional Near-Infrared Spectroscopy (fNIRS) is an alternative neuroimaging technique to fMRI that measures a similar physiological phenomenon. fNIRS uses specialized light emitting diodes that emit light in the near-infrared spectrum through the hair, scalp, skull, and meninges into the cortex. The light interacts with blood in the brain before refracting back to the surface where its intensity is measured by specialized photoreceptors. Due to subtle changes in the colour of blood depending on hemoglobin oxygenation status, the concentrations of oxygenated (HbO) and deoxygenated (HbR) hemoglobin can be inferred using the modified Beer-Lambert law. When a region of the brain becomes active, there is an initial dip in the concentration of HbO which is quickly met with an influx of oxygenated blood courtesy of neurovascular coupling. While this response can take up to ten seconds to peak, fNIRS is capable of sampling the cortex at 5Hz. In comparison to the typical sampling rate of 0.5Hz offered by fMRI, fNIRS offers superior temporal resolution. To reach the cortex and sample effectively, fNIRS detectors are typically placed about 3cm away from sources. Dense coverage provides a spatial resolution of about 1cm - ideal for studying cortical areas like the sensorimotor area. The NIRSport2 (NIRx Medical Technologies, LLC) is a portable system that is entirely contained in a small wearable pack. Compared to an fMRI machine, fNIRS is easier to use and more readily available. Additionally, there are no known contraindications to fNIRS, making it more useful for a clinical population who are ineligible to receive an MRI, enabling greater generalizability.

Taken together, generating an understanding of the neural mechanisms that allow cryoneurolysis to provide long-lasting spasticity relief using fNIRS and TMS will improve the understanding of the nature of recovery from spasticity, will potentially inform the clinical treatment of spasticity in the future, and may guide the development of future, brain-specific interventions for spasticity.

ELIGIBILITY:
Inclusion Criteria:

* are a patient at Parkwood Institute
* have increased range of motion or reduced spasticity with diagnostic nerve block,
* have no undesired loss of function with a diagnostic nerve block,
* score 2 or higher in the Modified Ashworth scale,
* have at least flickers of movement in the upper extremity,
* have not received botulinum-A neurotoxin within the past 3 months, and
* they can understand and follow instructions in English.

Exclusion Criteria:

* have contraindications to TMS (i.e., history of seizure, pregnancy) or 3T MRI (i.e., certain metallic implants),

  * are unable to provide informed consent (i.e., severe cognitive impairment),
  * receive any antispastic medication (oral, intrathecal, or otherwise) over the course of the follow-up period
  * receive any toxin injections for spasticity (Botulinum-A Toxin or equivalent) within 3 months of initial baseline assessments or at any time over the course of the follow-up period.
  * Have previously undergone any nerve-specific interventions (phenol neurolysis, radio-frequency ablation, or cryoneurolysis) for spasticity on a nerve that will be targeted for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
TMS | 6-months compared to baseline
  changes in cortical excitability
fNIRS | 6-months compared to baseline
  changes in hemoglobin concentration connectivity

SECONDARY OUTCOMES:
TMS | immediately post cryoneurolysis, 1-month post, 3-months post compared to baseline
  changes in cortical excitability
fNIRS | immediately post cryoneurolysis, 1-month post, 3-months post compared to baseline
  changes in hemoglobin concentration connectivity

OTHER OUTCOMES:
modified Ashworth Scale | change from baseline to 6 months
  Impairment measure - spasticity severity
Active range of motion | change from baseline to 6-months
  amount of movement
Modified Tardieu Scale | change from baseline to 6-months
  Impairment measure - spasticity severity/passive range of motion
Grip strength | change from baseline to 6-months
  Physical measurement - grip strength
EQ-5D-5L | change from baseline to 6-months
  health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sue Peters, PhD, Principal Investigator — Western University
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
With a low sample size (N=25) the risk of de-identification of participants is high. Summary statistics (e.g. mean) will be provided in the primary outcome manuscript.